CLINICAL TRIAL: NCT05140798
Title: Abu Dhabi Diabetes and Obesity Study -2 Bariatric
Acronym: ADOS-2B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IREC026
Record Dates: First submitted 2021-10-05; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric Surgery; Resting Metabolic Rate; Monogenic Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study on outcomes on bariatric surgery, particularly in terms of metabolic parameters in the UAE is scant. Also Genetic data from this population is limited and hence a study on genetic determinants of response to bariatric surgery is highly warranted. This study is expected to provide a better understanding of the causes of severe obesity in the UAE population and help us to evaluate the efficacy of Bariatric surgery in patients with genetic forms of obesity. The information generated will allow us to better advise patients regarding the risks and benefits of Bariatric Surgery as a treatment.

Objective To investigate the metabolic outcomes of bariatric surgery, to study the prevalence of monogenic forms of obesity among a cohort of patients with morbid obesity who underwent bariatric surgery and to compare the outcomes of Bariatric surgery in patients with and without underlying genetic condition.

DETAILED DESCRIPTION:
Prior to participation, the nature of the study, the objectives of the study, the study procedures and any known or likely risks including specific information pertaining to the genetic testing technology will be explained to the subjects by the study team.

Written informed consent will be obtained after providing an information sheet with details regarding the study including the genetic analysis performed. The information sheet with consent form will be available in Arabic and English. The participant (or parent/guardian or legally authorised representative, as appropriate) must personally sign and date the latest approved version of the ICF before any study specific procedures are performed.

A copy of the signed ICF will be kept in the medical record, with the study data, and provided to the participant. The original signed ICF will be retained at the study site for 10 years after the end of the project and should be conveyed to ICLDC, to be stored electronically, for its records.

Each subject will be informed that their source medical records may be checked by representatives from the responsible authorities (ICLDC REC, ADHRTC, DOH) with applicable regulations. However, they will be made aware that all information will be treated with confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending ICLDC who are planning to undergo, or who have already undergone BS for treatment of severe obesity.

Exclusion Criteria:

* Any malignant or chronic inflammatory disease,
* Children in the absence of parental consent
* Anyone who is not able to take part for reasons of significant incapacity or disability, including mental disability, preventing discussion of clinical history.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be patients attending ICLDC with severe obesity, who have previously had, or are considering metabolic surgery and also control group of patients who are not considering bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-04-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 3 months post BS
  Body composition including weightloss will be measured SECA body composition analyser
Change in weight | 6months post BS
  Body composition including weightloss will be measured SECA body composition analyser
Change in weight | 12months post BS
  Body composition including weightloss will be measured SECA body composition analyser
Change in weight | 18 months post BS
  Body composition including weightloss will be measured SECA body composition analyser
Change in weight | 24 months post BS
  Body composition including weightloss will be measured SECA body composition analyser
Change in weight | 36 months post BS
  Body composition including weightloss will be measured SECA body composition analyser
Change in resting metabolic rate | 3months post BS
  Our body uses energy while at rest, which we will be measuring it using an indirect calorimeter. The subject should ideally be fasting for at least 8 hrs before the procedure. If they are eligible, then they will asked to lie down on a couch with their upper body covered with a transparent hood, they will relax and breathe normally during the procedure .
Change in resting metabolic rate | 6 months post BS
  Our body uses energy while at rest, which we will be measuring it using an indirect calorimeter. The subject should ideally be fasting for at least 8 hrs before the procedure. If they are eligible, then they will asked to lie down on a couch with their upper body covered with a transparent hood, they will relax and breathe normally during the procedure .
Change in resting metabolic rate | 12 months post BS
  Our body uses energy while at rest, which we will be measuring it using an indirect calorimeter. The subject should ideally be fasting for at least 8 hrs before the procedure. If they are eligible, then they will asked to lie down on a couch with their upper body covered with a transparent hood, they will relax and breathe normally during the procedure .
Change in resting metabolic rate | 18 months post BS
  Our body uses energy while at rest, which we will be measuring it using an indirect calorimeter. The subject should ideally be fasting for at least 8 hrs before the procedure. If they are eligible, then they will asked to lie down on a couch with their upper body covered with a transparent hood, they will relax and breathe normally during the procedure .
Change in resting metabolic rate | 24 months post BS
  Our body uses energy while at rest, which we will be measuring it using an indirect calorimeter. The subject should ideally be fasting for at least 8 hrs before the procedure. If they are eligible, then they will asked to lie down on a couch with their upper body covered with a transparent hood, they will relax and breathe normally during the procedure .
Change in resting metabolic rate | 36 months post BS
  Our body uses energy while at rest, which we will be measuring it using an indirect calorimeter. The subject should ideally be fasting for at least 8 hrs before the procedure. If they are eligible, then they will asked to lie down on a couch with their upper body covered with a transparent hood, they will relax and breathe normally during the procedure .

SECONDARY OUTCOMES:
Change in liver fat | 3 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver fat. They may decide whether or not to consent.
Change in liver fat | 6 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver fat. They may decide whether or not to consent.
Change in liver fat | 12 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver fat. They may decide whether or not to consent.
Change in liver fat | 18 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver fat. They may decide whether or not to consent.
Change in liver fat | 24 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver fat. They may decide whether or not to consent.
Change in liver fat | 36 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver fat. They may decide whether or not to consent.
Change in liver thickness | 3 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver thickness. They may decide whether or not to consent.
Change in liver thickness | 6 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver thickness. They may decide whether or not to consent.
Change in liver thickness | 12 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver thickness. They may decide whether or not to consent.
Change in liver thickness | 18 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver thickness. They may decide whether or not to consent.
Change in liver thickness | 24 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver thickness. They may decide whether or not to consent.
Change in liver thickness | 36 months post BS
  If required, the subject may be asked to undergo an ultrasound elastography to analyse the liver thickness. They may decide whether or not to consent.
Change in serum leptin | 3 months post BS
  serum leptin
Change in serum leptin | 6 months post BS
  serum leptin
Change in serum leptin | 12 months post BS
  serum leptin
Change in serum leptin | 18 months post BS
  serum leptin
Change in serum leptin | 24 months post BS
  serum leptin
Change in serum leptin | 36 months post BS
  serum leptin
Change in insulin | 3 months post BS
  insulin
Change in insulin | 6 months post BS
  insulin
Change in insulin | 12 months post BS
  insulin
Change in insulin | 18 months post BS
  insulin
Change in insulin | 24 months post BS
  insulin
Change in insulin | 36 months post BS
  insulin
Change in serum cortisol | 3 months post BS
  serum cortisol
Change in serum cortisol | 6 months post BS
  serum cortisol
Change in serum cortisol | 12 months post BS
  serum cortisol
Change in serum cortisol | 18 months post BS
  serum cortisol
Change in serum cortisol | 24 months post BS
  serum cortisol
Change in serum cortisol | 36 months post BS
  serum cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Nader Lessan, MBBS MD FRCP CCST, Principal Investigator — Imperial College London Diabetes Centre
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided